CLINICAL TRIAL: NCT00930345
Title: A Study of Biological, Pathological and Imagery Markers in the First-line Treatment of Metastatic Clear-cell Renal Cell Carcinoma With Sunitinib BEFORE and AFTER Nephrectomy
Brief Title: Biological, Pathological and Imagery Markers in the First-line Treatment of Metastatic Clear-cell Renal Cell Carcinoma
Acronym: PREINSUT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070104
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2009-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Antiangiogenics; Biomarkers; Imagery
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SUTENT before nephrectomy (Other)
  Interventions: Drug: Sunitinib (SUTENT)

INTERVENTIONS:
Drug: Sunitinib (SUTENT) — Sunitinib, SUTENT, 50 mg daily p.o., on schedule 4/2, for 2 cycles. Two weeks of rest prior to surgery (week 11 and 12).
  Radical nephrectomy at the end of week 12. Sunitinib 50 mg/d, schedule 4/2, reintroduced 2 weeks after surgery (week 14, may be postponed by one or two weeks if wound healing delay or surgical complications). Treatment until disease progression, unacceptable toxicity or consent withdrawal. Dose reduction depending on the type and severity of toxicity.
  At the end of the treatment period patients will be treated at the discretion of the Investigator.

SUMMARY:
The aim of this study is to identify and/or validate biomarkers and imaging markers to predict and monitor the activity of a new class of therapeutic agents called antiangiogenics for the treatment of metastatic renal cell carcinoma (mRCC). Suntinib, approved for this indication, will be administred before and after nephrectomy and biomarkers sampling and imaging will be operated to monitor the activity and identify prognostic factors in mRCC.

DETAILED DESCRIPTION:
BACKGROUND Sunitinib, SUTENT, is a promising multi-target TKI in the treatment of metastatic renal cell carcinoma after cytokine failure. In previous phase II studies, ORR is 40% and TTP = 8,7 months. A phase III randomized trial of Sunitinib versus interferon alpha as first-line therapy for patients with mRCC showed a significantly longer PFS in the Sunitinib group (11 months) than in the interferon group (5 months), hazard ratio of 0.42 (95% CI, 0.32 to 0.54, p < 0.001). Initial approval in second line treatment of mRCC was extended to first line therapy on 11-01-2007.

Mechanisms of action involved in the therapeutic effects of antiangiogenic compounds are not fully elucidated. As of today, there are no validated biomarkers or imaging markers to predict and monitor the activity of this type of compound.

Recent findings in the field of cancer biology, tumor angiogenesis, immunology and imaging provide several biomarker candidates that can be assessed in metastatic renal cell carcinoma.

BASIC RESEARCH Biomarkers It seems interesting to measure the different biological markers that could be modulated by this antiangiogenic therapeutic. Some of them are known as prognostic factors in the metastatic renal carcinoma, others are directly linked to the mechanism of action of Sunitinib. Due to the biopsy prior to treatment initiation and nephrectomy after treatment initiation, it will be possible to evaluate biomarkers modification and to assess the potential link with the tumour response.

VHL gene alterations (mutations, deletions, and hypermethylations) are observed at high frequencies of up to 80% in cases of clear-cell renal cell carcinoma. The molecular mechanisms involved in angiogenesis in the presence of such genetic alterations are not yet well known. The functions of the pVHL/aHIF/VEGF/angiogenesis pathway will be investigated in all the renal cell carcinoma obtained from the biopsy and nephrectomy. Molecular markers defined by VHL status, expression and proteomic profiling may be helpful in predicting the responders.

Sunitinib is a potent inhibitor of the tyrosine kinase activity of several receptors: VEGFR-2, the main receptor responsible for mediating the proangiogenic effects of vascular endothelial growth factor (VEGF), expressed by vascular endothelial cells; PDGFR, the receptor for the platelet-derived growth factor (PDGF), expressed in pericytes which serve as structural supporting cells for endothelial cells. Consistent with its biochemical activity, Sunitinib inhibits the in vitro mitogenic response of human umbilical vein endothelial cells (HUVECs) stimulated by VEGF or bFGF (basic fibrosblast growth factor), another proangiogenic factor.

VEGF gene polymorphisms In physiologic and pathologic conditions, important variations in VEGF blood levels have been reported to correlate with constitutional VEGF-A gene polymorphisms located in intronic regions. Moreover, VEGF-A polymorphisms have been described as predisposition and prognostic factors in several human malignancies such as bladder, breast, melanoma, prostate and head and neck carcinomas. Hence, it is interesting to see whether these polymorphisms could affect tumor and clinical presentation and correlate with VEGF-levels and response to antiangiogenic treatment with sunitinib.

Immunology Tumor angiogenesis can impact immune response in renal cell carcinoma patients. A naturally occurring CD4+ T cell subset, regulatory CD4+CD25+ T cells, has emerged as the dominant T cell population governing peripheral self- tolerance by inhibiting effector T cell. The ability of anti-angiogenic therapy to block VEGF may allow better maturation of dendritic cells and a reduction of the number of regulatory CD4+CD25+T cells.

The aim of this project will be to test whether the administration of Sunitinib modulates the concentrations of regulatory CD4+CD25+T cells, and if a correlation between the immunology parameters and the response can be observed.

Imaging Radiological evaluation of tumor response is also challenging with anti-angiogenic drugs. Criteria based solely on size may be inadequate for evaluation of anti-angiogenic therapy efficacy. The unbridled expansion of tumor vessels leads to development of abnormal vessels, with distinct microvascular characteristics: high perfusion (blood flow), and porous walls leaking molecules into the interstitium (permeability).

New imaging techniques as dynamic contrast-enhanced CT are being developed to quantify and characterize these unique properties, and may be used as markers of response to angiogenesis inhibitors. Imaging assays of angiogenic status therefore offer the potential to clinically measure anti angiogenic effects of drugs on the tumor vessels themselves, effects that may not be reflected in changing tumor dimensions. These effects may be detectable hours or days from time of treatment initiation, rather than in weeks or months needed typically to detect a change in tumor size. Exploration of local tumor vascular architecture can help to understand mechanism of action of Sunitinib. This vasculature seems to be of poor functionality and tumor vascularization cannot be adequately assessed only by global index such as global tumor blood flow. In addition, exploration of renal tumor vascularization with contrast-enhanced US will be performed to compare blood flow determined by CT and US.

ELIGIBILITY:
Inclusion criteria :

* Patients with renal tumor in place, resectable, with at least one measurable metastasis 1.5 cm and indication of antiangiogenic therapy
* Histopathologically confirmed clear cell renal cell carcinoma (biopsy) and possibility of adequate tumor sampling prior to treatment
* No prior systemic treatment for RCC
* Male or female, 18 years
* Performance status ECOG 0-1
* Life expectancy 3 months
* Adequate organ function as defined by the following criteria:
* Total serum bilirubin 2 x ULN (Gilbert's disease exempt)
* Serum transaminases and alcalines phosphatases 2.5 x ULN, or in case of liver or bone metastasis 5x ULN

  * Serum creatinine 2 x ULN, creatinine clearance 80 ml/mn
  * Absolute neutrophil count (ANC) 1500/mm3
  * Platelets 100,000/mm3
  * Hemoglobin 10.0 g/dL
  * INR 1.7 or prothrobin time (PT) 6sec over
* Negative pregnancy test within 7 days prior to registration
* Signed and dated IRB/ICE-approved informed consent.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Patient covered by the national health system

Exclusion criteria :

* Previous nephrectomy
* Renal sarcoma, papillary tumors or collecting duct carcinoma
* Treatment in a clinical trial in the last 30 days
* Previous treatment with Sunitinib or other antiangiogenics
* Any of the following within 12 months prior to treatment initiation: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, thrombo-embolic accident or cerebrovascular accident including transient ischemic attack.
* Uncontrolled hypertension defined as systolic blood pressure >150mmHg or diastolic pressure >90mmHg, despite optimal medical treatment
* Ongoing cardiac dysrhythmia of grade 2, atrial fibrillation of any grade, QTc interval >0.50
* Treatment with anticoagulant agents and treatment with therapeutic doses of warfarin within 2 weeks prior to first day of Sunitinib. Low dose warfarin for deep vein thrombosis prophylaxis is permitted up to 2mg/day. Low molecular weight heparin or aspirin are allowed
* Any medical condition that might interfere with oral medication absorption
* Brain metastasis. Note: Brain scan or MRI is mandatory
* LVEF value < 50%
* Prior radiation therapy.
* Pregnancy or breastfeeding. Women and men must agree to use effective contraception during the study period. Acceptable contraception includes implants, oral contraceptives, intrauterine devices, surgical sterilization.
* Any acute or chronic medical or psychiatric condition or laboratory abnormality that would make the patient inappropriate with this study.
* Any second malignancy within the last 5 years with the exception of basal cell carcinoma, cervical cancer in situ and pT1/a bladder cancer with no evidence of recurrent disease for 12 months.
* Hypersensitivity to the Sunitinib malate or any excipient of Sutent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the prognostic value of several factors (biomarkers and imaging) to identify responders | 36 weeks

SECONDARY OUTCOMES:
To determine the objective response rate after initiation of treatment in the primitive tumour, according to the RECIST criteria. | 12 weeks
To assess the pathological response (tumoral extension), Progression Free Survival (PFS) as defined by pProgression Free Survival (PFS) as defined by progression of metastasis, overall survival (OS). | 24 months
To evaluate the correlation between tumor extension as defined by the pathologist and the tumor reduction between initiation of treatment and nephrectomy as measured by CT scan | 12 weeks
To compare marker expression in the biopsy (before treatment) and in the primitive tumor. | 12 weeks
To evaluate the ability of investigated biomarkers and VEGF-A gene polymorphisms to be prognostic of the pathological response and of the Progression Free Survival. | 24 months
To evaluate the correlation between the imaging obtained with Dynamic Contrast-enhanced CT scan, with contrast-enhanced US and VEGF expression | 6 weeks
To explore the pharmacokinetic of Sunitinib at study state | 4 weeks
To monitor the potential renal toxicity of Sunitinib | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephane OUDARD, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- HEGP, Paris, France